CLINICAL TRIAL: NCT05518162
Title: InBloom App vs ROSE Outcomes and Mechanisms
Brief Title: Treatment of Post-partum Depression Using an Behavioral Intervention Called ROSE (Reach Out, Stay Strong, Essentials for Mothers of Newborns) Delivered Using an Electronic App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen Poleshuck, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSRB00007456; R44MH112216 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Post-partum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- women receiving InBloom app (Experimental)
  Interventions: Device: InBloom
- women receiving ROSE as usual (Active Comparator)
  Interventions: Behavioral: ROSE
- historical controls- no treatment (No Intervention): We will capitalize on data from a large ROSE trial which consists of a demographically similar sample by comparing depression diagnosis outcomes for Inbloom and ROSE to the 96 participants in the care as usual group (an educational pamphlet on PPD).
- electronic health record utilization data (No Intervention): We will leverage EHR utilization data by retrospectively identifying 152 people from the same clinics who did not receive ROSE or InBloom and matched for eligibility criteria, demographics and PPD risk factors using propensity scores, and comparing their utilization to those in the ROSE and InBloom groups.

INTERVENTIONS:
Device: InBloom — The Rose Program (RPv2) application will be built for iOS and Android devices (including tablets) and will feature a video-based Learning Management System (LMS) which provides resources for people with postpartum depression to improve their wellbeing. Each InBloom session will contain 4-5 video modules with specific themes contained in each ROSE session which are 3-5 minutes each.
  Arms: women receiving InBloom app
Behavioral: ROSE — ROSE will be offered as a psychoeducational course on adjusting to parenthood by a health professional embedded in the obstetric clinics. There are five 90-minute group sessions which provide interpersonal rationale for the program, a review of the course outline, ground rules for the group, and the signs and symptoms of "baby blues" and postpartum depression, stress management skills. managing role transitions with an emphasis on transition to motherhood and the development of a support system, identifying types of interpersonal conflicts common around childbirth and techniques for resolving them, skills for resolving interpersonal conflicts and an opportunity to review and reinforce the content of the previous sessions.
  Arms: women receiving ROSE as usual

SUMMARY:
A randomized trial of pregnant people at risk for postpartum depression comparing the InBloom app (n = 76) to ROSE (n = 76; weekly scheduled group), and two control groups. We will assess Depression at baseline and 1, 2 and 3 months, ROI at 3 months, Satisfaction at 1 and 3 months and Perceived Access at 1 and 3 months. Subject participation will last up to 8 months (minimum 17 weeks pregnant through 3 months postpartum).

ELIGIBILITY:
Inclusion Criteria:

* 17-32 weeks pregnant
* enrolled for prenatal care in one of the five identified practices
* English speaking
* able to use an app (audio/visual/dexterity)
* have one or more of the following PPD risk factors: Medicaid eligible; anxiety (GAD-7 > 10) during pregnancy; mild to moderate depressive symptoms (PHQ-9 = 10-19); self-reported history of depression treatment; gestational diabetes; and/or young age (18-21 years).

Exclusion Criteria:

* patients with acute mental health needs
* cannot communicate in English
* demonstrate significant cognitive impairment
* are planning to place the child for adoption
* PHQ-9 depression score > 19
* younger than age 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of participants with post-partum depression assessed using the Mini International Neuropsychiatric Interview (MINI) | 3 months
  The MINI is a binary assessment of the diagnosis of postpartum depression. It yields a yes, no answer.
mean depression severity measured using Patient Health Questionnaire (PHQ-9) | baseline
  PHQ-9 is a 9 question tool that assesses depression symptoms. It ranges from 0-27 with higher scores indicating worse outcome.
mean depression severity measured using Patient Health Questionnaire (PHQ-9) | 1 month
  PHQ-9 is a 9 question tool that assesses depression symptoms. It ranges from 0-27 with higher scores indicating worse outcome.
mean depression severity measured using Patient Health Questionnaire (PHQ-9) | 2 months
  PHQ-9 is a 9 question tool that assesses depression symptoms. It ranges from 0-27 with higher scores indicating worse outcome.
mean depression severity measured using Patient Health Questionnaire (PHQ-9) | 3 months
  PHQ-9 is a 9 question tool that assesses depression symptoms. It ranges from 0-27 with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Return on Investment (ROI) | 3 months
  To calculate the return portion of ROI, all-cause healthcare utilization data of each patient will be obtained from the EHR. For each type of healthcare utilization, the corresponding per-unit reimbursement rate, obtained from New York State Medicaid fee schedule (https://omh.ny.gov/omhweb/medicaid_reimbursement/), which will then be multiplied by the utilization frequency to obtain the total reimbursement and thus total cost of care on a per-patient basis for each of the 3 groups. To calculate the investment portion of ROI, both the fixed costs (i.e., investment cost that does not vary by the number of patients treated) and the variable costs (i.e., investment cost that does vary by the number of patients treated) will be considered of the eROSE/ROSE intervention. Total utilization cost minus the intervention investment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Poleshuck E, Fox D, Abar B, Maeng D, Bilinski T, Beers L, Rosen J, Zlotnick C. Randomized clinical trial protocol of an app-based intervention to prevent postpartum depression. Contemp Clin Trials. 2025 Feb;149:107800. doi: 10.1016/j.cct.2024.107800. Epub 2024 Dec 30. PMID 39743016